CLINICAL TRIAL: NCT07282054
Title: A Phase 3, Randomized, Open-Label, Multicenter, Active-controlled Trial Comparing Efficacy and Safety of THDB0206 Injection With Insulin Lispro Injection Combined With Insulin Glargine Injection U-100 in Chinese Participants With Type 1 Diabetes
Brief Title: Efficacy and Safety of THDB0206 Compared to Insulin Lispro Injection in Participants With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tonghua Dongbao Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THDB0206L01
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THDB0206 Injection (Experimental)
  Interventions: Drug: THDB0206; Drug: Insulin Glargine
- Insulin Lispro Injection (Active Comparator)
  Interventions: Drug: Insulin Lispro; Drug: Insulin Glargine

INTERVENTIONS:
Drug: THDB0206 — Subcutaneous THDB0206 three times daily, with individualized dose adjustment.
  Arms: THDB0206 Injection
Drug: Insulin Lispro — Subcutaneous insulin lispro three times daily, with individualized dose adjustment.
  Arms: Insulin Lispro Injection
Drug: Insulin Glargine — Subcutaneous insulin glargine once daily, with individualized dose adjustment.

SUMMARY:
This is a 26-week randomized, open-label, multicenter, active-controlled parallel group trial. The purpose of this study is to compare efficacy and safety of THDB0206 injection with insulin lispro injection combined with insulin glargine injection U-100 in Chinese participants with T1DM.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, 18 to 75 years of age at informed consent (inclusive).
2. BMI between 18.0 and 30.0 kg/m² (inclusive).
3. T1DM diagnosed ≥6 months per WHO diabetes classification (2019).
4. On insulin therapy ≥6 months prior to screening.
5. Stable insulin regimen ≥3 months prior to screening (no change in insulin class), with or without metformin or alpha-glucosidase inhibitors; willing to follow multiple daily injections:

   1. Intermediate/long-acting insulin once or twice daily (e.g., NPH, glargine, detemir, degludec); plus prandial insulin 1~3 times daily (or as per usual diet) (e.g., regular human insulin, lispro, aspart, glulisine).
   2. Premixed insulin ≥2 times per day.
6. Screening HbA1c between 7.0% and 11.0% (inclusive), measured by the central laboratory.

Exclusion Criteria:

1. Diabetes other than T1DM.
2. History of pancreatectomy.
3. Prior pancreatic and/or islet cell transplantation.
4. ≥1 episode of Level 3 hypoglycemia within 6 months before screening (requires external assistance).
5. Hepatic or renal impairment at screening (per local laboratory reference ranges):

   1. AST or ALT ≥3× ULN; and/or
   2. TBL ≥2× ULN (except Gilbert syndrome); and/or
   3. Estimated creatinine clearance <45 mL/min (Cockcroft-Gault).
6. Known hypersensitivity/allergy to study insulin products or excipients, or to any component of the standardized test meal.
7. Blood transfusion or major blood loss within 3 months before screening; hemoglobinopathies, moderate-severe anemia, or other conditions that may interfere with HbA1c measurement.
8. Use of oral antihyperglycemics within 3 months before screening (except metformin and alpha-glucosidase inhibitors), or use of non-insulin injectables (e.g., GLP-1 receptor agonists).
9. Systemic corticosteroid therapy for ≥14 consecutive days within 3 months prior to screening (including IV, IM, SC, or oral routes; excluding topical, intraocular, intranasal, intra-articular, and inhaled use), or systemic corticosteroid therapy within 8 weeks prior to screening (except physiologic replacement for adrenal insufficiency), or anticipated need for prolonged systemic corticosteroid therapy during the study.
10. Use within 3 months before screening, or current use, of traditional medicines (herbal or proprietary Chinese medicines) with known glucose-lowering effects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in HbA1c at Week 26 | Week 26

SECONDARY OUTCOMES:
Change from Baseline in 1-hour Postprandial Glucose (PPG) Excursion at Week 26 | Week 26
Change from Baseline in 2-hour Postprandial Glucose (PPG) Excursion at Week 26 | Week 26

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: No